CLINICAL TRIAL: NCT03620903
Title: Efficacy of First Line Bortezomib, Rituximab, Ibrutinib (B-RI) for Patients With Treatment Naive Waldenström's Macroglobulinemia
Brief Title: Efficacy of First Line B-RI for Treatment Naive Waldenström's Macroglobulinemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Christian Buske (Other)
Collaborators: University of Ulm (Other); ClinAssess GmbH (Industry); Zentrum für Klinische Studien Ulm (Other); Hoffmann-La Roche (Industry); Johnson & Johnson (Industry)
Responsible Party: Sponsor-Investigator, Christian Buske, Prof. Dr. med., University of Ulm
Organization: University of Ulm (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECWM-2; 2017-004362-95 (EudraCT Number)
Record Dates: First submitted 2018-08-02; First posted 2018-08-08 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Waldenstrom Macroglobulinemia
Keywords: Waldenstrom Macroglobulinemia, Ibrutinib, Bortezomib
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — ibrutinib; Bortezomib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bortezomib-Rituximab-Ibrutinib (Experimental): Cycle 1:
  Rituximab: 375 mg/m2 intravenously (i.v) day 1; Bortezomib:1.6 mg/ m2 subcutanously (SC) day 1,8,15; Ibrutinib: 420 mg orally (p.o.) day 1-28;
  Cycle 2-6 Rituximab: 1400 mg absolute SC day 1; Bortezomib:1.6 mg/ m2 SC day 1,8,15; Ibrutinib: 420 mg p.o. day 1-28;
  Maintenance I (1 cycle = 56 days):
  Ibrutinib 420 mg p.o. daily, until evidence of progressive disease or no longer tolerated by the subject (for a maximum of 10 years); Rituximab 1400 mg absolute SC day 1, every second month for 24 months (month 7-30);
  Maintenance II (1 cycle = 84 days):
  Ibrutinib 420 mg p.o. daily, until evidence of progressive disease or no longer tolerated by the subject (for a maximum of 10 years);
  Interventions: Drug: Ibrutinib / Bortezomib / Rituximab

INTERVENTIONS:
Drug: Ibrutinib / Bortezomib / Rituximab — Induction (Rituximab / Bortezomib / Ibrutinib), Maintenance I (Ibrutinib / Rituximab), Maintenance II (Ibrutinib)
  Other Names: Imbruvica / Velcade / Mabthera

SUMMARY:
In Waldenström macroglobulinemia (WM) conventional chemotherapy induces only low complete remission (CR) rates and responses of short duration compared to other indolent lymphomas. Thus innovative approaches are needed which combine excellent activity and tolerability in patients with WM, who are mostly of advanced age. The immunochemotherapy DRC (dexamethasone, rituximab, cyclophosphamide) was shown to be highly effective in patients with WM without inducing major hematological toxicities. On the other hand the proteasome inhibitor bortezomib showed substantial activity as a single agent in WM with only very few side effects when given in a weekly schedule. Recent data confirmed high activity with low toxicity for ibrutinib in relapsed WM patients as single agent therapy. Based on these observations it is the aim of this study to investigate the efficacy and toxicity of the chemotherapy-free combination bortezomib, rituximab, ibrutinib (B-RI) in treatment naïve WM patient.

DETAILED DESCRIPTION:
In Waldenström's macroglobulinemia (WM) conventional chemotherapy induces only low complete remission (CR) rates and responses of short duration compared to other indolent lymphomas. Thus innovative approaches are needed which combine excellent activity and tolerability in patients with WM, who are mostly of advanced age. Today, chemotherapy in combination with the anti-cluster of differentiation (CD) 20 antibody rituximab is still the backbone of treatment in patients with WM and is recommended as first line in national and international treatment guidelines. With the approval of Ibrutinib by the European Medicines Agency (EMA) 2015 for patients with relapsed WM or for patients not eligible for chemotherapy with treatment naïve WM treatment landscape has changed in this lymphoma subtype and there is an urgent need to evaluate to which extent chemotherapy-free approaches add clinical benefit to the patient. The treatment in the "European Consortium for Waldenström's Macroglobulinemia" (ECWM)-2 trial will test, whether the chemotherapy-free approach, which is given orally (ibrutinib) and subcutaneously (bortezomib and rituximab from cycle 2 onwards) (B-RI) will approach the efficacy of chemotherapy containing treatment concepts, but avoids chemotherapy associated toxicity. From the perspective of single agent ibrutinib, this regimen tests whether ibrutinib can be further optimized by adding rituximab and bortezomib. The combination of rituximab and ibrutinib was tested in comparison to rituximab/placebo in a large international phase III trial on behalf of the European Consortium for Waldenström's Macroglobulinemia in relapsed and first line WM, and results were recently published: in this trial no unexpected toxicity of the combination ibrutinib/rituximab was reported. Furthermore, ibrutinib/rituximab was significantly superior to rituximab/placebo with regard to response rates and PFS. From the perspective of the established rituximab/bortezomib regimen, the combination of B-RI will evaluate whether adding ibrutinib to this combination will add any benefit for the patient.

To this end, the aim of the study is to assess the toxicity and efficacy of B-RI in an exploratory phase II trial.

ELIGIBILITY:
Inclusion Criteria

* Clinicopathological diagnosis of WM as defined by consensus panel one of the Second International Workshop on WM, diagnosed by a reference pathology center. Pathological diagnosis has to occur before study inclusion. In addition, pathological specimens have to be sent to the national pathological reference center at study inclusion. The positivity for Cluster of Differentiation (CD) 20 can be assumed from any previous bone marrow immunohistochemistry or flow cytometry analysis performed up to 6 months prior to enrollment. Inclusion in the study will be based on morphological and immunological criteria. Immunophenotyping will be performed in each center and saved locally. Flow cytometry of bone marrow and blood cells will include at least one double staining and assess the expression of the following antigens: surface immunoglobulin, CD19, CD20, CD5, CD10 and CD23. Patients are eligible if tumor cells express the following antigens: CD19, CD20, and if they are negative for CD5, CD10 and CD23 expression. Patients with tumor cells positive for CD5 and/or CD23 and morphologically similar to WM cells may be included after ruling out other low-grade B-cell malignancies.
* Presence of at least one criterion for initiation of therapy, according to the 2nd Workshop on WM:

  * Recurrent fever, night sweats, weight loss, fatigue (at least one of them)
  * Hyperviscosity
  * Lymphadenopathy which is either symptomatic or bulky (≥5 cm in maximum diameter)
  * Symptomatic hepatomegaly and/or splenomegaly
  * Symptomatic organomegaly and/or organ or tissue infiltration
  * Peripheral neuropathy due to WM
  * Symptomatic cryoglobulinemia
  * Cold agglutinin anemia
  * Immunoglobulin M (IgM) related immune hemolytic anemia and/or thrombocytopenia
  * Nephropathy related to WM
  * Amyloidosis related to WM
  * Hemoglobin ≤10g/dL
  * Platelet count <100x109/L
  * Serum monoclonal protein >5g/dL, even with no overt clinical symptoms
* Low or absent IgG serum levels
* World Health Organization (WHO)/Eastern Co-operative Oncology Group (ECOG) performance status 0 to 2.
* Other criteria:

  * Age ≥ than 18 years
  * Life expectancy >3 months.
  * Baseline platelet count >100x10exponential (E)9/L if not due to bone marrow (BM) involvement by the lymphoma, independent of any transfusions
  * absolute neutrophil count >1x10E9/L independent of growth factor support.
  * Meet the following pretreatment laboratory criteria at the Screening visit conducted within 28 days of study enrollment:

    * aspartate aminotransferase (AST): <3 times the upper limit of institutional laboratory normal value
    * alanine aminotransferase (ALAT): <3 times the upper limit of institutional laboratory normal value
    * Total Bilirubin: < 1.5 times the upper limit of institutional laboratory normal value, unless clearly related to the disease (except if due to Gilbert's syndrome)
    * Serum creatinine: ≤ 2 times the upper limit of institutional laboratory normal value or estimated Glomerular Filtration Rate (cockroft-gault ≥ 40 mL/min/1.73m2)
* Premenopausal fertile females must agree to use a highly effective method of birth control for the duration of the therapy up to 6 months after end of therapy. A highly effective method of birth control is defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomised partner.
* Men must agree not to father a child for the duration of therapy and 12 months after and must agree to advice a female partner to use a highly effective method of birth control.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Affiliation to a social security scheme (relevant for France only)

Exclusion Criteria:

* Prior systemic treatment of the WM (plasmapheresis and short - term administration of corticosteroids < 4 weeks administered at a dose equivalent to < 20 mg/day prednisone is allowed)
* Patient with hypersensitivity to Bortezomib
* Patient with hypersensitivity to MabThera
* Patient with hypersensitivity to Ibrutinib
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Uncontrolled viral infection
* Known history of human immunodeficiency virus (HIV) or active Hepatitis C Virus or active Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (IV) antibiotics.
* Congenital or acquired severe immunodeficiency not attributed to lymphoma (clinical appearance: recurrent infections, necessity of immunoglobulin substitution therapy, patients after transplantation)
* Known interstitial lung disease
* Prior allergic reaction or severe anaphylactic reaction related to humanized or murine monoclonal antibody.
* Central Nervous System involvement by lymphoma
* Prior history of malignancies unless the subject has been free of the disease for ≥ 5 years. Exceptions include the following:
* Basal cell carcinoma of the skin,
* Squamous cell carcinoma of the skin,
* Carcinoma in situ of the cervix,
* Carcinoma in situ of the breast,
* Incidental histologic finding of prostate cancer (TNM stage of T1a or T1b).
* Uncontrolled illness including, but not limited to:
* Uncontrolled diabetes mellitus (as indicated by metabolic derangements and/or severe diabetes mellitus related uncontrolled organ complications)
* Chronic symptomatic congestive heart failure (Class New York Heart Association (NYHA) III or IV).
* Unstable angina pectoris, angioplasty, stenting, or myocardial infarction within 6 months
* Clinically significant cardiac arrhythmia that is symptomatic or requires treatment, or asymptomatic sustained ventricular tachycardia.
* Known pericardial disease
* acute diffuse infiltrative pulmonary and pericardial disease
* Subjects with ≥ Grade 2 neuropathy.
* Recent major surgery (within 4 weeks prior to study inclusion)
* History of stroke or intracranial haemorrhage within 6 months prior to study inclusion
* Women who are pregnant as well as women who are breast-feeding and do not consent to discontinue breast-feeding.
* Participation in another clinical trial within four weeks prior to study inclusion
* No consent for registration, storage and processing of the individual disease-characteristics and course as well as information of the family physician about study participation
* St. John's Wort with Ibrutinib
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon).
* Requires treatment with strong cytochrome P (CYP) 3A inhibitors.
* Vaccinated with live, attenuated vaccines within 4 weeks prior to study inclusion.
* Person of legal age who is incapable of comprehending the nature, significance and implications of the clinical trial and of determining his/her will in the light of these facts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
1 year progression free survival | 1 year
  The primary endpoint is the rate of 1 year progression free survival (1YPFS).

SECONDARY OUTCOMES:
Response rate | 6 months
  response rates (CR, VGPR, PR, MR) and overall response rate (CR, VGPR, PR, MR)
Best response | up to 10 years
  At least achieving a MR
Time to best response | up to 10 years
  time from the start of induction to best response the patient achieves (CR, VGPR, PR, MR).
Time to first response | up to 10 years
  time from the start of induction to first response (MR, PR, VGPR or CR).
Time to Treatment failure (TTF) | up to 10 years
  time of start of induction treatment to discontinuation of therapy for any reason including death from any cause, progression, toxicity or add-on of new anti-cancer therapy.
Remission duration (RD) | up to 10 years
  patients with response (CR, VGPR, PR, MR) from the date of response to the date of progression, relapse or death from any cause.
Progression Free Survival (PFS) | up to 10 years
  date of start of treatment to the following events: the date of progression and the date of death if it occurred earlier.
Cause specific survival (CSS) | up to 10 years
  period from the start of induction treatment to death from lymphoma or lymphoma related cause
Overall survival (OS) | up to 10 years
  period from the start of induction treatment to death from any cause.
Safety Analysis | up to 10 years
  Safety including treatment associated adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Buske, MD, Principal Investigator — University of Ulm
Locations (12):
- Germany (11):
  - Studiengesellschaft Onkologie Bielefeld GbR, Bielefeld
  - DIAKO Ev. Diakonie-Krankenhaus gGmbH, Med. Klinik II, Bremen
  - Universitätsklinikum Halle, Klinik für Innere Medizin IV, Halle
  - Universtätsmedizin Mannheim, III. Medizinische Klinik Studienzentrale im MCC, Mannheim
  - Kliniken Maria Hilf GmbH (Krankenhaus St. Franziskus), Medizinische Klinik I (Klinik f. Hämatologie, Onkologie, Gastroentereologie), Mönchengladbach
  - Kliniken Ostalb Stauferklinikum Schwäbisch Gmünd, Zentrum für Innere Medizin, Mutlangen
  - Hämato-Onkologische Gemeinschaftspraxis Pasing-Fürstenfeldbruck, München
  - Klinikum der Universität München, Medizinische Klinik und Poliklinik III, München
  - Universitätsklinikum Münster, Med. Klinik A, Münster
  - Universitätsklinikum Ulm; Klinik für Innere Medizin Innere Medizin III, Ulm
  - Gemeinschaftspraxis Dres. Rudolf Schlag, Björn Schöttker, Joachim Haas, Würzburg
- 'Alexandra' General Hospital of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: No